CLINICAL TRIAL: NCT00239876
Title: A Two-year Extension to a One-year, Multicenter, Open-label, Randomised Study to Evaluate the Safety and Efficacy of FTY720 Combined With Tacrolimus and Steroids Versus Mycophenolate Mofetyl Combined With Tacrolimus and Steroids, in de Novo Adult Renal Transplant Recipients
Brief Title: Efficacy and Safety of FTY720 in de Novo Adult Renal Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720A2302E1
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Renal Transplantation
Keywords: Transplantation, kidney, and organ transplant
MeSH Terms: interventions — Fingolimod Hydrochloride

INTERVENTIONS:
Drug: FTY720

SUMMARY:
This study will evaluate the safety and efficacy of FTY720 combined with tacrolimus and corticosteroids in patients receiving a kidney transplant

ELIGIBILITY:
Inclusion Criteria

* Completed the 12 month core study
* Informed consent Exclusion Criteria
* N/A Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2005-05; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
IA, IB, IIA, IIB, III, or humoral rejection diagnosed by biopsy according to Banff 97 criteria within 36 months post transplant
Permanent resumption of dialysis within 36 months post transplant
Surgical removal of graft within 36 months post transplant
Death within 36 months post transplant
Withdrawal of consent, death, or lost to follow up within 36 months post transplant
Serum creatinine, estimated creatinine clearance, assessment of other laboratory abnormalities and vital signs and measurement of urine protein. at Months 18, 24, 30 and 36
Pulmonary FEV1 , FVC, FEV1/FVC, DLCO and FEF 25%-75% at Months 18, 24, 30 and 36
Absolute lymphocyte count at Month 18, 24, 30 and 36.

SECONDARY OUTCOMES:
Physical examinations at Months 18, 24, 30 and 36
Vital signs at Months 18, 24, 30 and 36
Electrocardiogram at Months 24 and 36
Chest X-ray Months 24 and 36
Safety laboratory tests 18, 24, 30 and 36
Ophthalmic evaluations 18, 24, 30 and 36
AEs and SAEs
FTY720/CsA levels at Months 18, 24, 30 and 36

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis